CLINICAL TRIAL: NCT03086317
Title: USAT-CDT Trial: Standard vs Ultrasound-assisted Catheter Thrombolysis for Submassive Pulmonary Embolism
Brief Title: Standard vs Ultrasound-assisted Catheter Thrombolysis for Submassive Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Wissam Jaber, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00093040
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Diseases
Keywords: Pulmonary Medicine; Therapy Evaluation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two treatments for acute, submassive pulmonary embolism.
Who Masked: Outcomes Assessor
Masking Description: Pre- and post-treatment computed tomography angiography (CTA) will be compared by independent radiologists who are blinded to the type treatment received.
  Pre- and post-treatment echocardiograms will be interpreted by independent cardiologists who are blinded to the type of treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Catheter-Directed Thrombolysis (Active Comparator): Participants randomized to this arm will receive standard catheter-directed thrombolysis, per standard of care, as treatment for acute submassive pulmonary embolism.
  Interventions: Device: Standard Catheter-Directed Thrombolysis
- Ultrasound-Accelerated Thrombolysis (Active Comparator): Participants randomized to this arm will receive ultrasound-accelerated thrombolysis, per standard of care, as treatment for acute submassive pulmonary embolism.
  Interventions: Device: Ultrasound-Accelerated Thrombolysis

INTERVENTIONS:
Device: Standard Catheter-Directed Thrombolysis — Catheter-directed thrombolysis requires placement of a multi-sidehole infusion catheter within the pulmonary arterial thrombus burden, under angiographic guidance. Thrombolytic medications are slowly infused through the catheter, which is left in place for the duration of the treatment. The treatment will be performed according to current standard of care and all technical considerations will be left to the discretion of the operator performing the procedure. All follow up is according to standard of care.
  Other Names: CDT
  Arms: Standard Catheter-Directed Thrombolysis
Device: Ultrasound-Accelerated Thrombolysis — USAT is a modification of standard catheter-directed thrombolysis utilizing a proprietary system of local high frequency, low-power ultrasound to dissociate the fibrin matrix of the thrombus, allowing deeper penetration of lytic medication. The treatment will be performed according to current standard of care and all technical considerations will be left to the discretion of the operator performing the procedure. All follow up is according to standard of care.
  Other Names: USAT
  Arms: Ultrasound-Accelerated Thrombolysis

SUMMARY:
The study is an investigator-initiated trial comparing two different catheters (standard versus ultrasound assisted) for the treatment of acute high risk pulmonary embolism (blood clots in lung arteries with evidence or heart strain). Patients already planned for the procedure will be randomized to standard catheter-directed thrombolysis (CDT) or to ultrasound-assisted catheter thrombolysis (USAT). Both catheters are currently used routinely in practice for the treatment of pulmonary embolism, but it is not known if USAT is superior to standard CDT, the former being much more expensive and more commonly used.

The purpose of the study is to learn about which catheter-directed therapy is more suitable for patients with pulmonary embolism (PE), who are candidates for both standard catheter directed therapy (CDT), and ultrasound-assisted catheter directed therapy (USAT), and to provide information regarding the cost effectiveness of the two different types of treatment. A total of 80 patients are planned to be recruited. All medication administration, procedures or in-hospital tests will be performed as routine clinical practice. The study will compare short term and long term outcomes: resolution of blood clots on CT scan, right ventricular size improvement, quality of life and symptoms at 3 and 12 months, and cost effectiveness.

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) accounts for 5-10% of in-hospital deaths. Systemic anticoagulation (AC) is the standard of care and thrombolysis is recommended for those at a higher mortality risk. Catheter-directed therapies, mainly standard catheter-directed thrombolysis (CDT) and ultrasound-accelerated thrombolysis (USAT), have been introduced as new, more effective, and safer treatment modalities. USAT is a modification of standard catheter thrombolysis, utilizing a system of local ultrasound to dissociate the fibrin matrix of the thrombus, allowing deeper penetration of lytics. However, there is limited data comparing the two treatments. More rapid clearance of pulmonary thrombus by USAT compared to standard CDT may prove to be more effective regarding clinical outcomes and cost (e.g. via reduced length of ICU and hospital stay). Alternatively, if thrombus clearance is similar, the cost of USAT may exceed the cost of CDT (equipment and disposables), without offering any potential advantage.

This controlled, randomized study seeks to determine if ultrasound acceleration adds any benefits in the outcomes and costs of catheter-directed thrombolysis for patients with acute submassive PE. The treatment with CDT or USAT are standard of care for submassive PE and participants will be randomized to receive one treatment or the other. Participants will have follow up visits at 3 months and 12 months post procedure. All the procedures, tests, and follow up visits are according to current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for catheter directed thrombolysis per the study protocol for submassive pulmonary embolism (PE)

  * CT or echocardiographic RV strain (defined as RV/LV ratio >1)
  * without persisting hypotension <90mmHg or drop of systolic blood pressure by at least 40mm Hg for at least 15 minutes with signs of end-organ hypoperfusion (cold extremities or low urinary output <30 mL/h or mental confusion)
* without the need of catecholamine support
* without the need of cardiopulmonary resuscitation

Exclusion Criteria:

* Pregnancy
* Index PE symptom duration >14 days
* High bleeding risk (any prior intracranial hemorrhage, known structural intracranial cerebrovascular disease or neoplasm, ischemic stroke within 3 months, suspected aortic dissection, active bleeding or bleeding diathesis, recent spinal or cranial/brain surgery, recent closed-head or facial trauma with bony fracture or brain injury)
* Participation in any other investigational drug or device study
* Life expectancy <90 days
* Inability to comply with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Jaber, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Health System and Emory Healthcare System in Atlanta, Georgia, USA. Participant enrollment began October 19, 2017, and all follow-ups were completed by December 8, 2020.
Period: Overall Study
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10) | 43 (15) | 50 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18
Concomitant Deep Venous Thrombosis [Count of Participants; unit: Participants] | 3 | 5 | 8
Mean Oxygen at Baseline [Number; unit: percentage of oxygen saturation] | 92 | 95 | 94
Mean Heart Rate (HR) at baseline [Number; unit: beats per minute] | 98 | 106 | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Thrombus Obstruction
Description: Computed tomography angiography (CTA) will be performed before and after treatment. An independent radiologist will quantify the degree of obstruction from the thrombus by determining the vascular obstruction index. For determining the CT obstruction index, the arterial tree of each lung will be considered to have 10 segmental arteries (three to the upper lobes, two to both the middle lobe and the lingula, and five to the lower lobes).
Time Frame: Baseline to end of lysis treatment (up to 72 hours)
Measure: Mean (Standard Deviation); unit: percentage of thrombus obstruction
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
percentage of thrombus obstruction
  Baseline ratio | 33 (4) | 31 (4)
  End of lysis treatment (up to 72 hrs) | 23 (7) | 22 (7)

2. Secondary Outcome: In Hospital Mortality
Description: Mortality during hospitalization will be compared between the two study arms.
Time Frame: Until hospital discharge (an average of 6 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

3. Secondary Outcome: 90-day Mortality
Description: Mortality until 90 days post procedure will be compared between the two study arms.
Time Frame: Until 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

4. Secondary Outcome: Cardiac Decompensation Due to Massive Pulmonary Embolism
Description: Cardiac decompensation, defined as hypotension (<90 millimeters of mercury (mmHg)) and use of catecholamines, will be compared between the two study arms.
Time Frame: Through follow up (12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

5. Secondary Outcome: Major Bleeding
Description: Major bleeding is defined as overt bleeding associated with a hemoglobin level reduction of at least 2.0 grams per deciliter (g/dL), or with transfusion of two or more units of red blood cells, or involvement of a critical site (intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome).
Time Frame: Through follow up (12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

6. Secondary Outcome: Minor Bleeding
Description: Clinically overt bleeding not fulfilling the criteria of major bleeding is classified as a minor bleeding complication.
Time Frame: Through follow up (12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Participants | 0 | 1

7. Secondary Outcome: Symptomatic Venous Thromboembolism (VTE)
Description: Recurrent venous thromboembolism (VTE) will be diagnosed if symptoms or signs of deep vein thrombosis or acute pulmonary embolism (PE) are confirmed by an imaging test. There will be no routine surveillance for asymptomatic recurrent VTE.
Time Frame: Until 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

8. Secondary Outcome: Clinical Success of Treatment
Description: Treatment will be considered successful if pulmonary embolism related decompensation is prevented, without the participant experiencing a major adverse event or death.
Time Frame: Until 90 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Participants | 10 | 8

9. Secondary Outcome: ICU Length of Stay
Description: The number of days participants were admitted to the ICU will be compared between study arms.
Time Frame: Until hospital discharge (an average of 6 days)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
Days | 2 [2 to 5] | 2 [1 to 58]

10. Secondary Outcome: Change in Right Ventricular/Left Ventricular (RV/LV) Diameter Ratio
Description: Under normal circumstances, the right ventricle appears smaller than the left ventricle when measured by an echocardiogram (RV/LV ratio<1). An increased RV/LV ratio may be a predictor of poor clinical outcomes following pulmonary embolism.
Time Frame: Baseline, end of lysis treatment, Month 3, Month 12
Population: Endpoint results include only participants who showed up for the study visits.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
ratio
  Baseline (RV/LV) diameter ratio | 1.7 (0.4) | 1.5 (0.3)
  End of Lysis Treatment (RV/LV) diameter ratio | 1.1 (0.2) | 1.2 (0.2)
  Month 3: number analyzed (Participants) | 10 | 5
  Month 3 | 0.87 (0.3) | 0.89 (0.2)
  Month 12: number analyzed (Participants) | 6 | 6
  Month 12 | 0.82 (0.2) | 0.84 (0.2)

11. Secondary Outcome: Change in Tricuspid Annular Plane Systolic Excursion (TAPSE)
Description: Tricuspid annular plane systolic excursion (TAPSE) is an echocardiographic of measuring right ventricular function. TAPSE measurements can be categorized as normal (1.5-2.0cm), mildly abnormal (1.3-1.5cm), moderately abnormal (1.0-1.2cm) or severely abnormal (<1.0cm).
Time Frame: Baseline, end of lysis treatment, Month 3, Month 12
Population: Data was not collected
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Right Ventricular Systolic Pressure (RVSP)
Description: Right ventricular systolic pressure (RVSP) measured by echocardiogram provides an estimate the pressure inside the artery supplying blood to the lungs. Dysfunction in the right ventricle is assessed to predict clinical outcomes following pulmonary embolism.
Time Frame: Baseline, end of lysis treatment, Month 3, Month 12
Population: Results reflect participants who completed study procedures during each study visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 10 | 8
mmHg
  Baseline | 55 (14) | 50 (10)
  End of lysis Treatment: number analyzed (Participants) | 2 | 2
  End of lysis Treatment | 42 (0) | 38 (0)
  Month 3: number analyzed (Participants) | 8 | 4
  Month 3 | 36 (12) | 37 (19)
  Month 12: number analyzed (Participants) | 4 | 4
  Month 12 | 32 (10) | 34 (16)

13. Secondary Outcome: Number of Participants Who Had a Decrease in New York Heart Association (NYHA) Functional Classification of Heart Failure From Class 4 to Class 2
Description: New York Heart Association (NYHA) Functional Classification of heart failure classifies heart failure with a combination of two methods: patient symptoms and objective assessment by a healthcare provider. Patient symptoms are classified as I-IV, where I = "no limitation of physical activity" and IV = "unable to carry on any physical activity without discomfort". An objective assessment by a healthcare provider is classified as A through D where A = "objective evidence of cardiovascular disease" and D = "objective evidence of severe cardiovascular disease".
Time Frame: Month 3, Month 12
Population: All participants had a baseline NYHA Class 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 6 | 5
Participants
  Month 3- Number of participants with NYHA Class 2 | 2 | 2
  Month 12: number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in 6-minute Walk Test
Description: The 6-minute walk test (6MWT) measures the distance that can be quickly walked by the study participant in 6 minutes. A 30 meter long walking course is created using cones on a hard, flat surface and the participant will walk the course as many times as they can in 6 minutes while a study team member counts the number of laps completed. Specific test guidelines from the American Thoracic Society will be followed.
Time Frame: Month 3, Month 12
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 7 | 2
meters
  Month 3 | 360 (131) | 330 (28)
  Month 12 | 336 (14) | 387 (92)

15. Secondary Outcome: Change in 36-Item, Short Form (SF-36) Score
Description: The SF-36 is a 36 item survey assessing the quality of life across the 8 domains of physical functioning, limitations due to physical health, limitations due to emotional health, energy, emotional well-being, social functioning, pain, and general health. Each item is scored between 0 and 100 where 0 represents the worst possible quality of life and 100 corresponds with a healthy state of being. The numbers analyzed below represent the average score obtained with 0 being the bottom 25% of the quality of life (score 0-25), 1 is 26-50, 2 is 51-75, and 4 is 76-100.
Time Frame: Month 3, Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 7 | 5
score on a scale
  Month 3 | 3.1 (0.94) | 3.17 (0.69)
  Month 12 | 3.43 (0.73) | 3.6 (0.49)

16. Secondary Outcome: Change in Quality of Life After Pulmonary Embolism (PEmb QoL) Score
Description: Quality of life after pulmonary embolism (PEmb QoL) questionnaire is a 40 item survey asking respondents about their lung symptoms after having a pulmonary embolism. Participants report on 6 dimensions which cover the frequency and intensity of lung symptoms, physical and social limitations due to symptoms, pain, and emotional distress following having a pulmonary embolism. Scoring the responses involves specific instructions to reverse the scores for several dimensions, resulting in a score between 0 and 100 where 0 corresponds with "no complaints" and 100 is "worst possible" outcome.
Time Frame: Month 3, Month 12
Population: Data not collected
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change in Shortness of Breath Questionnaire Score
Description: The University of California San Diego (UCSD) Medical Center Shortness of Breath Questionnaire is a 24 item survey asking respondents how much shortness of breath they experience doing particular activities. Breathlessness is rated on a scale of 0 (not at all breathless) to 5 (maximally breathless or unable to do an activity become of breathlessness). Total scores range from 0 to 120, with higher scores indicating increased shortness of breath.
Time Frame: Month 3, Month 12
Population: Data was not collected
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Cost Effectiveness Analysis
Description: A Markov state-transition, cost effectiveness model will be created to simulate patient oriented outcomes assuming a societal perspective with a 12-month time horizon. All point estimates for model parameters will be determined from the prospectively collected data. Quality adjusted life years will be determined for each therapy based on survival, freedom from major adverse events, discharge status, functional status, and quality of life measures. Costs will be calculated for each therapy based on in-hospital resource utilization (i.e., length of stay in the ICU, operating room and procedure costs, and associated adverse event costs) and out-of-hospital costs (outpatient nursing care, loss of work, outpatient testing and follow-up).
Time Frame: Month 12
Population: Data was not collected
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning after randomization up to 90 days after randomization.
Arm/Group | Standard Catheter-Directed Thrombolysis | Ultrasound-Accelerated Thrombolysis
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03086317/Prot_SAP_000.pdf